CLINICAL TRIAL: NCT04477005
Title: Prospective Observational Cohort Study: To Assess the Utility of Bio-degradable Bile Duct Stent in the Drainage of Bile Duct.
Brief Title: Archimedes Bio-degradable Bile Duct Stent Study
Acronym: ABBS
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20GA041
Record Dates: First submitted 2020-06-26; First posted 2020-07-20 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Bile Leak; Common Bile Duct Stone With Chronic Cholecystitis
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ERCP and insertion ofBio-degradable bile duct stent — ERCP is an accepted mode of treatment and patients rarely need surgery for bile leaks and bile duct stents. Endoscopic management involves sphincterotomy (cutting open the Sphincter of Oddi) and insertion of a plastic or metal stent. Instead of placing a plastic stent bio-degradable stent will be placed. They will be followed up on Day 1, 7,30, 60,90 and 180 days. they will have abdominal x-ray on day 90 and day180.
  Other Names: Archimedes BD stent

SUMMARY:
This is a prospective observational cohort study to assess the utility of bio-degradable bile duct stent in the drainage of bile duct. All consecutive patients who will undergo ERCP procedure for bile leaks and patients with bile duct stones and intact gall bladder will be recruited to the study. The planned sample size is 53 and patients will be followed up for 180 days. The primary objective is to assess the utility of biodegradable bile duct plastic stents in the drainage of bile duct.

The secondary Secondary objectives are To assess

1. Technical success of biodegradable stents
2. Complications
3. Patient related cost savings (Time off work, travel time for the patient)
4. Hospital related cost savings (Repeat procedure costs, follow up appointments)

DETAILED DESCRIPTION:
This is a Multi-centre prospective observational cohort study assessing biodegradable stents in the drainage of bile duct. The participating organisations are Nottingham university hospitals NHS trust which is the host and sponsor of this study, University college London Hospitals NHS foundation trust and Leeds teaching hospitals NHS trust.

The population studied will be patients who need temporary bile duct stent insertion for bile leak and patients who had ERCP for removal of CBD stones and have stones either in the neck of gall bladder or cystic duct and awaiting cholecystectomy. These are the group of patients who may not benefit from a repeat endoscopic procedure to remove the stent. As the target population is rare, all consecutive patients with above condition will be recruited to the study.

All patients who are referred for ERCP will be screened to see if they meet the eligibility criteria to participate in the study. The patient information sheet (PIS) will be sent to the patient along with the endoscopy appointment. The pateints will be consented both for the procedure and the study on the day of the procedure. Then the patients will have the procedure in their respective endoscopic units. All ERCP procedures will be done either by an accredited endoscopist or by a trainee under the close supervision of the accredited endoscopist.

Once the patients have their treatment, the patients will be observed for four hours for complications. Then discharged home if they are well and do not have any symptoms such as pain, persistent low blood pressure (defined as systolic less than 100) and have recovered from the effects of sedation. If at all the pateints develop any of the above symptoms, then the patients will be admitted for an overnight observation. The patients will have a telephone consultation by research specialist nurses the next day to assess if they have symptoms such as abdominal pain, vomiting, vomiting of blood and dark tarry stools. If the patients develop any of these symptoms, the patients will be assessed in the bio-medical research centre or respective inpatient facility in relevant centres. The patients will then have a blood test including full blood count, liver function and renal function. Amylase will be done only if they complain of abdominal pain as a proportion of patients will have hyper-amylasaemia following ERCP. The patients will also receive a telephone consultation (Research nurse) on day 7 post procedure to assess if they have any of the above symptoms. A quality of life questionnaire will be completed at this stage.

The investigators will be using slow degrading stents so, therefore the patients will have an abdominal x-ray 90 days after the procedure and if the stent is not visible on abdominal X-ray then they would have completed the study. As recent studies have shown that the stent appear partially degraded in some patients, if the stent is visible on x-ray then the patients will have one more follow up visit with an abdominal x-ray at 180 days. The invetstigator will not remove the stent as the stent would have partially degraded and would have lost its tensile strength.

Almost all bile leaks are inpatients so the resolution of bile leak will be assessed while they are inpatients. The resolution of bile leak is defined as no output from the external drain that was inserted through the skin under radiological guidance. For bile duct stones it is the prevention of bile duct infection (Cholangitis). The pateints will have telephone consultations on days 1,30,60,90 and 180 to asses if they have symptoms such as abdominal pain, jaundice. A quality of life questionnaire (EQ-5D-5L) will be completed at all these visits. Once the patient completes all of the above, they will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study.

  * Male or Female, aged 18 years or above.
  * Patients who have an indication for ERCP.
  * Patients who have bile leak either post cholecystectomy or liver resection.
  * Patients who are on the waiting list for cholecystectomy for gall stones but have bile duct stones and listed for removal of bile duct stones.
  * Able (in the Investigators opinion) and willing to comply with all study requirements.
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Female participants who is pregnant, lactating or planning pregnancy during the course of the study.
* Patients who are unable to consent for the study.
* Participant who is terminally ill
* Patients who come for ERCP and routine stent change
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who need ERCP for bile leak or bile duct stones except participants who are pregnant or breast feeding.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Resolution of bile leak | 180 days
  In patients who have bile leak post HPB surgery, They will have an external drain to drain the leaked bile. Resolution of bile leak is defined as no output of bile through the external drain.
Incidence of cholangitis in patients who had ERCP for bile duct stones and are awaiting gall bladder removal. | 180 days
  Cholangitis- infection of bile duct ( fever, rigors, elevated white cell count and CRP). Incidence of cholangitis post procedure will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Vasan Venkatachalapathy, MRCP(Gastr), Principal Investigator — NIHR Nottingham BRC,Nottingham University Hospitals NHS Trust and the University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All personal identifiable information collected during the study will be coded, depersonalised with unique codes for each patient. The study will be compliant with the requirements of the General Data Protection Regulation 2018 and the Data Protection Act 2018.
  The CRF will only collect the minimum required information for the purposes of the trial. CRFs will be held securely, in a locked room in a locked cupboard.All patient data will be stored in an encrypted computer with password access at the NIHR Nottingham BRC, Nottingham University Hospitals NHS Trust and the University of Nottingham. Members other than the direct care team will not have access to this data.